CLINICAL TRIAL: NCT06878248
Title: A Phase 1, Open-Label, Dose-Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Combination of CLBR001, an Engineered Autologous T Cell Product, and ABBV-461, an Antibody-Based Biologic, in Subjects With Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study to Assess CLBR001+ABBV-461 in Subjects With Locally Advanced or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBR-sCAR461-3001
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Metastatic; Locally Advanced Breast Cancer (LABC); Malignant Neoplasm of Breast; Triple Negative Breast Cancer (TNBC); Hormone Receptor-Positive Breast Cancer; HER2 + Breast Cancer
Keywords: breast cancer; CAR-T therapy; metastatic breast cancer; locally advanced breast cancer; malignant neoplasm of breast; Triple Negative Breast Cancer; hormone receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Combination product CLBR001 + ABBV461 is administered in ascending dose level cohorts to determine the Optimal Biologic Dose (OBD) of CLBR001 + ABBV-461.
  Interventions: Biological: Two Component Product CLBR001 + ABBV-461

INTERVENTIONS:
Biological: Two Component Product CLBR001 + ABBV-461 — Investigational switchable CAR-T cell therapy for breast cancer

SUMMARY:
The goal of this clinical trial is to evaluate CLBR001 and ABBV-461 as a treatment for patients with locally advanced or metastatic breast cancer. The goals are to establish the safety and efficacy of the combination therapy while establishing the optimal biologic doses.

Patients will be administered a single infusion of CLBR001 cells followed by cycles of ABBV-461 with regular assessments of safety and disease response to treatment.

DETAILED DESCRIPTION:
CLBR001 + ABBV-461 is novel switchable CAR-T cell combination therapy comprised of an autologous CAR-T product (CLBR001, the switchable CAR-T cell [sCAR-T]) and ABBV-461 (the "switch" biologic molecule). ABBV-461 acts as an adapter molecule that controls the activity of the CLBR001 CAR-T cell product.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed locally advanced or metastatic breast cancer
* Exhaused all standard of care therapy options
* Measurable disease at time of screening in accordance with RECIST v1.1 criteria
* Women or men age ≥18 years of age at time of consent
* ECOG performance status 0 or 1
* Must provide a biopsy sample obtained during the screening period, following the end of the most recent prior line of therapy
* Adequate hematological, renal, and liver function

Exclusion Criteria:

* History of a clinically significant infection within 4 weeks prior to consent
* Active bacterial, viral, and/or fungal infection
* Prior allogeneic stem cell transplant
* Prior lentiviral- or retroviral-based therapy including CAR-T cell therapy
* Prior lymphodepleting or T-cell cytotoxic therapy within 3 months of enrollment
* Subjects receiving attenuated vaccines within 4 weeks of consent or need for live vaccine within 12 months of starting study therapy
* History of significant cardiovascular conditions within the past 6 months
* Subjects with a prior history of or concurrent malignancy whose natural history or treatment has the potential to interfere with either the safety or efficacy assessment of the investigational regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events as assessed by CTCAE v5.0 and ASTCT consensus grading criteria for CRS and ICANS | To 1-year post administration of CLBR001
  To assess the safety and tolerability in subjects by evaluating the frequency, relatedness, severity and duration of adverse events, as assessed by CTCAE v5.0 and ASTCT consensus grading criteria for CRS and ICANS.
Number of subjects with replication competent lentivirus | To 1-year post administration of CLBR001
  To assess the safety and tolerability in subjects by evaluating the number of subjects testing positive for replication competent lentivirus.
Number of dose-limiting toxicities as assessed by CTCAE v5.0 and ASTCT consensus grading for CRS and ICANS | To 28-days post-first dose of ABBV-461
  The number of dose-limiting toxicities as assessed by CTCAE v5.0 and ASTCT consensus grading for CRS and ICANS will be used to identify an Optimal Biologic Dose (OBD) of CLBR001 and ABBV-461.

SECONDARY OUTCOMES:
Pharmacodynamics | To 1-year post administration of CLBR001
  To measure pharmacodynamic response by evaluating concentrations of serum cytokines.
Assess Immunogenicity using Antidrug Antibodies | To 1-year post administration of CLBR001
  To determine Immunogenic response to CLBR001 and ABBV-461 by presence of antidrug antibodies (ADA)
Overall Best Objective Response | To 1-year post administration of CLBR001
  To evaluate anti-tumor activity of CLBR001 + ABBV-461 by assessing Overall (best) objective response by response evaluation criteria in solid tumors by using RECIST v1.1.
Disease Control Rate | To 1-year post administration of CLBR001
  To evaluate anti-tumor activity of CLBR001 + ABBV-461 by assessing Disease Control Rate by using RECIST v1.1.
Evaluate Pharmacokinetics of CLBR001 + ABBV-461 : Cmax | To 1-year post administration of CLBR001
  To evaluate the pharmacokinetics (PK) of CLBR001, including expansion and persistence, and ABBV-461 by quantifying CLBR001 cells in peripheral blood and PK parameters of ABBV-461.
Evaluate Pharmacokinetics of CLBR001 + ABBV-461 : Tmax | To 1-year post administration of CLBR001
  To evaluate the pharmacokinetics (PK) of CLBR001, including expansion and persistence, and ABBV-461 by quantifying CLBR001 cells in peripheral blood and PK parameters of ABBV-461.
Evaluate Pharmacokinetics of CLBR001 + ABBV-461 : AUC | To 1-year post administration of CLBR001
  To evaluate the pharmacokinetics (PK) of CLBR001, including expansion and persistence, and ABBV-461 by quantifying CLBR001 cells in peripheral blood and PK parameters of ABBV-461.
Evaluate Pharmacokinetics of CLBR001 + ABBV-461 : t(1/2) | To 1-year post administration of CLBR001
  To evaluate the pharmacokinetics (PK) of CLBR001, including expansion and persistence, and ABBV-461 by quantifying CLBR001 cells in peripheral blood and PK parameters of ABBV-461.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Study Director — Calibr-Skaggs Institute for Innovative Medicines
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No